CLINICAL TRIAL: NCT03337711
Title: A Open Multicenter Clinical Study to Explore Intra-tumor Heterogeneity and Prognostic Value of Postoperative Blood ctDNA of ⅡA - ⅢA Stage Non-squamous NSCLC Based on the Capture-based Sequencing and UMI (Unique Molecular Identifier) Technology of Burning Rock
Brief Title: Explore Intra-tumor Heterogeneity and Prognostic Value of Postoperative Blood ctDNA of ⅡA - ⅢA Stage Non-squamous NSCLC Based on the Capture-based Sequencing and UMI Technology of Burning Rock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hao Long, professor, Sun Yat-sen University
Other Study IDs: A2017-001
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC;ctDNA;IIA-IIIA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The relationship of postoperative ctDNA and recurrence defined by clinical imaging will be analyzed, as well as the correlation of tissue and postoperative blood NGS results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will collect 100 ⅡA - ⅢA stage non-squamous NSCLC tumor tissue and blood specimens (Include: (1) tissue by operation: 3 specimens from different regions of each patient; (2) Blood: preoperative blood (within one week), postoperative blood (3-4 weeks after operation (before adjuvant chemotherapy), 20 weeks after operation (1 month after adjuvant chemotherapy), 1 year after operation). Capture-based sequencing(168 genes panel +UMI) will performed. All patients are recommended for "pemetrexed combined platinum" adjuvant chemotherapy for 4 cycles(Moderate-dose Chemotherapy) 3-4 weeks after operation. The clinical data should be collected until disease progression. The relationship of postoperative ctDNA and recurrence defined by clinical imaging will be analyzed, as well as the correlation of tissue and postoperative blood NGS results.

ELIGIBILITY:
Inclusion Criteria:

1. Received radical surgical treatment and postoperative pathological had pointed out non-squamous NSCLC;
2. Patients with postoperative pathologic staging diagnosis of Ⅱ A - Ⅲ A period (AJCC TNM staging (version 8));
3. Female or male Age ≥ 18 years and ≤ 75;
4. Did not receive any of the anti-tumor treatment for current disease, such as radiation therapy, chemotherapy, or molecular target, etc;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0/1；
6. The expect survival time is more than 6 months;
7. Screening laboratory results:

(1) Hematological:Absolute Neutrophil Count (ANC) ≥ 1500 K/mm^3 (without use of G-CSF 4 weeks prior to enrollment);Hemoglobin (Hgb) ≥ 9 g/dL (transfusions allowed);Platelets (Plts) ≥ 100 k/mm^3; (2) Hepatic:Bilirubin ≤1.5×upper limit of normal (ULN),Aspartate aminotransferase (AST) ≤2.5 × ULN, ≤ 5 x ULN if liver metastases are present;Alanine aminotransferase (ALT) ≤ 2.5 × ULN, ≤ 5 x ULN if liver metastases are present; (3) Renal:Cr≤ 1.5 x ULN or Ccr≥ 50 mL/min, and Urine dipstick test result show urinary protein < 2+. The urinary protein ≥ 2 + should be 24-hour urine collection and ensure 24 hours urine protein content < 1 g; 8. Patients agreed and have the ability to follow the study plan to be visited, agreed to provide blood specimens in the process of preoperative (within one week) and postoperative (3-4 weeks, 20 weeks and 1 year after surgery) and tumor tissue specimens by operation, and cooperate with other research steps.

Exclusion Criteria:

1. Second primary malignancy, other than cervical carcinoma in situ after adequate treatment, in situ malignancies or adequately treated basal cell carcinoma of the skin, localized prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery;
2. Clinical evaluation for patients with inoperable;
3. A serious uncontrolled medical disorder or active infection that in the investigator's opinion would impair the participant's ability to receive study treatment;
4. Prior therapy with surgery, chemotherapy, targeted therapy and immunotherapy is not allowed;
5. Eastern Cooperative Oncology Group performance status(ECOG PS ) ≥2;
6. A definite clinical active infection, including but not limited to pneumonia;
7. Other situation the researchers think that doesn't fit into the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postoperative pathologic staging diagnosis of ⅡA to ⅢA non-squamous NSCLC period
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
recurrence or metastasis | two years after the last patient entered the study
  The patient was diagnosed as recurrence or metastasis according to the computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided